CLINICAL TRIAL: NCT01045993
Title: A Pilot Study To Evaluate Various Methodologies For Assessing The Treatment Of Low Back Pain
Brief Title: A Study To Evaluate Methods To Evaluate Back Pain
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Wyeth is now a wholly owned subsidiary of Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: TC-09-20
Record Dates: First submitted 2010-01-08; First posted 2010-01-11 (Estimated); Results first posted 2013-04-01 (Estimated); Last update posted 2013-04-01 (Estimated); Status verified 2013-02

CONDITIONS: Pain
Keywords: Pilot Study to Assess Methodologies
MeSH Terms: conditions — Pain

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No

ARMS (4):
- 1 (Active Comparator): Heat device
  Interventions: Device: Heat Device
- 2 (Sham Comparator): Placebo arm
  Interventions: Device: Sham Device
- 3 (Active Comparator): Marketed analgesic
  Interventions: Drug: marketed analgesic
- 4 (Placebo Comparator): (Oral) Placebo comparator
  Interventions: Drug: Placebo

INTERVENTIONS:
Device: Heat Device — 8-Hour Heatwrap
  Other Names: Heatwrap
  Arms: 1
Device: Sham Device — Inactive wrap worn for 8 hours
  Arms: 2
Drug: marketed analgesic — 2 x 200 mg ibuprofen tablets
  Arms: 3
Drug: Placebo — 2 x placebo tablets
  Arms: 4

SUMMARY:
The study is designed to assess methods used in clinical research.

ELIGIBILITY:
Inclusion Criteria:

* Lower back pain
* Male or female in generally good health, from 18 to 55 years of age (inclusive)

Exclusion Criteria:

* Pregnant or lactating
* Subject has evidence or history of radiculopathy, i.e. sciatica extending below the knee (numbness, tingling, or shooting pain), or other neurologic deficits (abnormal straight leg raise test, patellar reflexes, and/or bowel and bladder function);
* Subject has a history of previous back surgery;
* Subject has back pain resulting from traumatic injury involving physical evidence of bruising, swelling, or inflammation to the abdomen or low back area which occurred less than 48 hours prior to enrollment
* Has taken an investigational drug within the past 30 days prior to entering the study, or currently enrolled in another investigational study
* Is a member or relative of the study site staff, CRO or Sponsor organization directly involved with the study or had a household member or relative participate concurrently or previously in this study
* Has previously been enrolled in this study

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 61 (Actual)
Dates: Start 2010-02; Primary Completion 2010-07 (Actual); Study Completion 2010-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (1):
- Pfizer Investigational Site, Loma Linda, California, United States

REFERENCES:
- [Derived] Stark J, Petrofsky J, Berk L, Bains G, Chen S, Doyle G. Continuous low-level heatwrap therapy relieves low back pain and reduces muscle stiffness. Phys Sportsmed. 2014 Nov;42(4):39-48. doi: 10.3810/psm.2014.11.2090. PMID 25419887
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=TC-09-20&StudyName=A%20Study%20To%20Evaluate%20Methods%20To%20Evaluate%20Back%20Pain

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were recruited who had primary muscular low back pain (in the Investigator's best judgment), which was atraumatic (no traumatic injury within 48 hours of enrollment) and not caused by, or related to, any clinically significant, medical diseases, whose onset had occurred within the past 3 months.
Pre-assignment Details: Eligible participants with at least moderate pain intensity on a 6-point categorical scale were randomized (N=61) to primary efficacy (heatwrap or oral placebo) or blinding groups ("sham" wrap or oral Ibuprofen). May have received rescue medication (oral acetaminophen) during the 4-hour evaluation period or at discharge after assessments completed.
Groups:
- ThermaCare®: Active treatment low back/hip heatwrap administered one time (could be applied for up to 8 hours); applied within 5 minutes of unsealing the foil wrapper.
- Sham Wrap (Inactive): Inactive heatwrap administered one time as a non-heating wrap; applied within 5 minutes of unsealing the foil wrapper.
- Oral Ibuprofen (IBU): IBU (commercially available Advil®) administered as two 200 milligram (mg) tablets by mouth (PO) as a one time dose.
- Oral Placebo: Oral Placebo matching Oral IBU.
Period: Overall Study
Arm/Group | ThermaCare® | Sham Wrap (Inactive) | Oral Ibuprofen (IBU) | Oral Placebo
Started | 26 | 5 | 5 | 25
Completed | 26 | 4 | 5 | 25
Not Completed | 0 | 1 | 0 | 0
Not completed — Treated-later found eligibility not met | 0 | 1 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | ThermaCare® | Sham Wrap (Inactive) | Oral Ibuprofen (IBU) | Oral Placebo | Total
Number analyzed (Participants) | 26 | 5 | 5 | 25 | 61
Age Continuous [Mean (Standard Deviation); unit: years] | 30.0 (6.0) | 25.6 (5.4) | 30.0 (7.2) | 28.8 (7.7) | 29.1 (6.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 11 | 1 | 2 | 15 | 29
  Male | 15 | 4 | 3 | 10 | 32
Number of participants with categorical score for pain intensity [Number; unit: participants] — Participant rated the severity of their pain on a 6-point scale in response to the question "How much pain are you experiencing in your lower back right now". Scored as None=0, Mild=1, Moderate=2, Moderately severe=3, Severe=4, Extreme=5. Participant was asked to remember the level of pain experienced at this time as a reference for any pain relief experienced at later time points.
  participants
    None=0 | 0 | 0 | 0 | 0 | 0
    Mild=1 | 0 | 0 | 0 | 0 | 0
    Moderate=2 | 19 | 3 | 2 | 20 | 44
    Moderately severe=3 | 7 | 1 | 3 | 4 | 15
    Severe=4 | 0 | 1 | 0 | 1 | 2
    Extreme=5 | 0 | 0 | 0 | 0 | 0
Back Stiffness Score [Mean (Standard Deviation); unit: millimeters] — Participant rated their low back muscle stiffness by placing a line on a visual analog scale (VAS) in response to the question "Please indicate a number from 0 through 100 that best describes your low back muscle stiffness". VAS scaled as 0 millimeters (mm) to 100 mm in length with 0 (no muscle stiffness) up to 100 (most possible stiffness).
  millimeters | 45.85 (13.18) | 55.00 (18.71) | 50.00 (10.61) | 51.24 (20.32) | 49.15 (16.67)
Flexibility Assessment: Extension (Angle) [Mean (Standard Deviation); unit: degree of angle] — Flexibility assessed using Paris Plinth table with maximum extension (as if performing a sit-up) of 20 degrees movement. Angle at baseline standardized to 100 for assessment of maximum angle (x degrees) up to the degree of movement at which participant perceives discomfort or pain, x degrees minus 5, and x degrees plus 5. Greater degree of angle indicated greater flexibility.
  degree of angle
    Maximum degrees | 15.31 (4.53) | 16.48 (4.82) | 16.80 (3.89) | 14.07 (4.51) | 15.02 (4.48)
    Minus 5 degrees | 10.19 (4.38) | 11.26 (5.04) | 11.62 (3.70) | 9.01 (4.28) | 9.91 (4.32)
    Plus 5 degrees (beyond maximum) | 17.28 (4.48) | 18.50 (2.24) | 18.78 (4.35) | 17.59 (4.02) | 17.63 (4.08)
Flexibility Assessment: Extension (visual analog scale ([VAS]) [Mean (Standard Deviation); unit: millimeters] — Flexibility assessed using Paris Plinth table with maximum extension (as if performing a sit-up) of 20 degrees movement. When participant feels discomfort or pain, participant places a mark to rate discomfort/pain on a VAS of 100 mm in length with 0=no discomfort/no pain up to 100=most discomfort/most pain. Movement decreased 5 degrees and discomfort rated on VAS. Movement increased 5 degrees beyond first point when pain was reported and discomfort/pain again rated on the VAS. Higher scores indicated greater pain.
  millimeters
    VAS at Maximum degrees | 48.65 (15.69) | 41.00 (21.21) | 48.20 (13.52) | 43.40 (23.35) | 45.84 (19.26)
    VAS at Minus 5 degrees | 33.54 (19.41) | 26.60 (22.00) | 34.00 (11.51) | 29.36 (22.37) | 31.30 (20.11)
    VAS at Plus 5 degrees (beyond maximum) | 56.92 (20.27) | 50.00 (32.64) | 59.40 (14.28) | 52.60 (27.47) | 54.79 (23.78)
Flexibility Assessment: Side-to-Side (Angle) [Mean (Standard Deviation); unit: degree of angle] — Flexibility assessed using Paris Plinth table with maximum side-to-side movement of plus or minus 10 degrees for left (L), and right (R), movement. Angle at baseline standardized to 100 for assessment of maximum angle (x degrees) up to the degree of movement at which participant perceives discomfort or pain, x degrees minus 5, and x degrees plus 5. Greater degree of angle indicated greater flexibility.
  degree of angle
    L Maximum degrees | 6.92 (1.69) | 7.20 (1.79) | 6.50 (2.40) | 7.16 (1.50) | 7.01 (1.65)
    R Maximum degrees | 6.80 (1.76) | 7.40 (1.34) | 6.50 (2.06) | 6.76 (1.80) | 6.81 (1.74)
    L Minus 5 degrees | 2.15 (1.19) | 2.40 (1.34) | 2.00 (1.41) | 2.32 (1.07) | 2.23 (1.15)
    R Minus 5 degrees | 2.05 (1.27) | 2.40 (1.34) | 1.80 (1.64) | 1.92 (1.19) | 2.00 (1.25)
    L Plus 5 degrees (beyond maximum) | 7.22 (1.66) | 7.40 (1.34) | 6.60 (2.19) | 7.42 (1.40) | 7.26 (1.56)
    R Plus 5 degrees (beyond maximum) | 7.33 (1.41) | 7.70 (0.67) | 7.00 (1.39) | 7.02 (1.68) | 7.20 (1.47)
Flexibility Assessment: Side-to-side (VAS) [Mean (Standard Deviation); unit: millimeters] — Flexibility assessed using Paris Plinth table with maximum side-to-side movement of plus or minus 10 degrees for left, and right, movement. When participant feels discomfort or pain, participant places a mark to rate discomfort/pain on a VAS of 100 mm in length with 0=no discomfort/no pain up to 100=most discomfort/most pain. Movement decreased 5 degrees and discomfort rated on VAS. Movement increased 5 degrees beyond first point when pain was reported and discomfort/pain again rated on the VAS. Higher scores indicated greater pain.
  millimeters
    L VAS at Maximum degrees | 42.69 (22.61) | 32.40 (14.64) | 43.60 (21.28) | 35.24 (25.87) | 38.87 (23.29)
    R VAS at Maximum degrees | 47.38 (25.18) | 40.40 (20.97) | 52.20 (14.45) | 45.40 (20.69) | 46.39 (22.03)
    L VAS at Minus 5 degrees | 24.85 (22.82) | 15.20 (9.47) | 28.20 (14.46) | 22.80 (18.77) | 23.49 (19.66)
    R VAS at Minus 5 degrees | 24.35 (19.57) | 19.80 (13.92) | 34.00 (19.96) | 24.96 (18.75) | 25.02 (18.68)
    L VAS at Plus 5 degrees (beyond maximum) | 40.58 (26.10) | 27.80 (15.42) | 48.20 (22.83) | 37.64 (25.93) | 38.95 (24.95)
    R VAS at Plus 5 degrees (beyond maximum) | 48.42 (26.16) | 42.40 (22.03) | 55.60 (13.63) | 44.92 (21.85) | 47.08 (23.05)
Flexibility Assessment: Rotation (Angle) [Mean (Standard Deviation); unit: degree of angle] — Flexibility assessed using Paris Plinth table with maximum rotation at waist movement of plus or minus 30 degrees for left, and right, movement. Angle at baseline standardized to 100 for assessment of maximum angle (x degrees) up to the degree of movement at which participant perceives discomfort or pain, x degrees minus 5, and x degrees plus 5. Greater degree of angle indicated greater flexibility.
  degree of angle
    L Maximum degrees | 15.67 (4.08) | 17.36 (3.77) | 15.96 (6.44) | 17.03 (4.40) | 16.39 (4.35)
    R Maximum degrees | 16.78 (4.73) | 16.66 (4.26) | 16.62 (6.19) | 16.91 (4.78) | 16.81 (4.71)
    L Minus 5 degrees | 10.21 (4.12) | 11.30 (4.09) | 10.42 (6.19) | 11.46 (4.33) | 10.83 (4.31)
    R Minus 5 degrees | 11.27 (4.48) | 11.28 (4.38) | 10.74 (6.12) | 11.56 (4.46) | 11.34 (4.49)
    L Plus 5 degrees (beyond maximum) | 17.95 (3.28) | 17.66 (3.73) | 17.12 (5.13) | 18.24 (4.12) | 17.98 (3.75)
    R Plus 5 degrees (beyond maximum) | 18.48 (4.14) | 18.46 (3.73) | 18.06 (4.39) | 18.32 (4.30) | 18.38 (4.10)
Flexibility Assessment: Rotation (VAS) [Mean (Standard Deviation); unit: millimeters] — Flexibility assessed using Paris Plinth table with maximum rotation at waist of plus or minus 30 degrees for left, and right, movement. When participant feels discomfort or pain, participant places a mark to rate discomfort/pain on a VAS of 100 mm in length with 0=no discomfort/no pain up to 100=most discomfort/most pain. Movement decreased 5 degrees and discomfort rated on VAS. Movement increased 5 degrees beyond first point when pain was reported and discomfort/pain again rated on the VAS. Higher scores indicated greater pain.
  millimeters
    L VAS at Maximum degrees | 52.54 (23.88) | 60.00 (23.74) | 60.60 (12.30) | 48.80 (23.41) | 52.28 (22.81)
    R VAS at Maximum degrees | 51.65 (21.33) | 59.40 (31.09) | 61.60 (15.84) | 49.64 (25.97) | 52.28 (23.56)
    L VAS at Minus 5 degrees | 36.92 (21.25) | 47.20 (22.94) | 46.60 (21.24) | 33.24 (22.28) | 37.05 (21.77)
    R VAS at Minus 5 degrees | 38.15 (22.26) | 44.20 (27.47) | 47.40 (15.84) | 36.56 (25.02) | 38.75 (23.12)
    L VAS at Plus 5 degrees (beyond maximum) | 56.62 (25.62) | 63.80 (18.79) | 65.80 (12.19) | 49.24 (22.12) | 54.93 (23.10)
    R VAS at Plus 5 degrees (beyond maximum) | 59.12 (27.10) | 66.40 (28.17) | 64.20 (11.50) | 50.92 (26.61) | 56.77 (26.08)

OUTCOME MEASURES:

1. Secondary Outcome: Time to Meaningful Relief
Description: Time to "meaningful relief" defined as elapsed time from start of treatment until participant depressed the second stopwatch indicating "meaningful relief" (meaningful to participant). Participant consider censored if participant did not depress the stopwatch by end of 4-hour in-patient evaluation, or became a treatment failure (rescue or discontinuation) during the time prior to depressing the second stopwatch. Censoring was at time of dropout if participant withdrew for non-efficacy related reasons during the 4-hour in-patient portion of the study. CI calculated using method of Simon & Lee.
Time Frame: Baseline (time of wrap application or oral treatment administration) up to 4 hours
Population: ITT population. Median and/or upper limit of CI reported as 240 minutes if median or upper limit >240 minutes.
Measure: Median (95% Confidence Interval); unit: minutes
Arm/Group | ThermaCare® | Sham Wrap (Inactive) | Oral Ibuprofen (IBU) | Oral Placebo
Number analyzed (Participants) | 26 | 5 | 5 | 25
minutes | 215.7 [163.7 to 240] | 104.0 [71.0 to 240] | 135.1 [119.8 to 240] | 240 [NA to NA] — CI was not calculated as time to meaningful pain relief was >240 minutes.
Statistical Analysis 1: Comparison: ThermaCare® vs Oral Placebo; Test type: Superiority or Other; p = 0.046, Proportional hazards regression model — Statistically significant treatment difference was declared if the probability of random occurrence between the treatment groups p-value was ≤0.05; P-value calculated using proportional hazards model with treatment term only in the model

2. Primary Outcome: Time to First Perceptible Relief (Confirmed by Meaningful Relief)
Description: "First perceptible relief" defined as the elapsed time from wrap application or oral treatment until the participant depressed the first stopwatch labeled "first perceptible relief" (any pain relieving effect), provided the participant also depressed the second stopwatch labeled "meaningful relief" (meaningful to participant) by the end of the scheduled in-patient evaluation (4 hours / 240 minutes). If the confirmation was not achieved, the participant was censored at the time when the first stopwatch was depressed. Confidence interval (CI) calculated using the method of Simon & Lee.
Time Frame: Baseline (time of wrap application or oral treatment administration) up to 4 hours
Population: Intent-to-treat population (ITT): all randomized participants who applied/dosed with study product and had a baseline assessment. Median and/or upper limit of CI reported as 240 minutes if >240 minutes. No primary endpoint was prespecified in this Pilot study; 1 key efficacy endpoint was selected for reporting purposes only.
Measure: Median (95% Confidence Interval); unit: minutes
Arm/Group | ThermaCare® | Sham Wrap (Inactive) | Oral Ibuprofen (IBU) | Oral Placebo
Number analyzed (Participants) | 26 | 5 | 5 | 25
minutes | 96.5 [26.4 to 240] | 38.7 [7.5 to 240] | 54.0 [31.3 to 240] | 240 [NA to NA] — CI was not calculated as time to first perceptible pain relief was >240 minutes.
Statistical Analysis 1: Comparison: ThermaCare® vs Oral Placebo; Test type: Non-Inferiority or Equivalence — The statistical alternative hypothesis tested is that the survival curves of time to first perceptible relief confirmed by meaningful relief are not identical between two treatment groups, or equivalently, the hazard ratio between two treatment groups is not equal to 1; p = 0.046, Proportional hazards regression model — [p-value comment as in outcome 1, analysis 1]; P-value calculated using proportional hazards model with treatment term only in the model

3. Secondary Outcome: Time Weighted Sum of Pain Relief From 0 Through 8 Hours (TOTPAR 0-8)
Description: TOTPAR 0-8 sum of pain relief from 0 through 8 hours, weighted by the time duration between the current timepoint and the previous timepoint. Pain relief rated hourly (from baseline) by the participant on a 6-point scale: 0=no relief, 1=a little relief, 2=less than half relief, 3=more than half relief, 4=a lot of relief, 5=complete relief. Total possible score 0 to 40; higher score indicated better relief.
Time Frame: Baseline (time of wrap application or oral treatment administration) up to 8 hours
Population: ITT population.
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | ThermaCare® | Sham Wrap (Inactive) | Oral Ibuprofen (IBU) | Oral Placebo
Number analyzed (Participants) | 26 | 5 | 5 | 25
scores on a scale | 22.0 (7.9) | 15.6 (13.1) | 17.0 (13.5) | 11.5 (10.0)
Statistical Analysis 1: Comparison: ThermaCare® vs Oral Placebo; Test type: Superiority or Other; p < 0.001, ANOVA — [p-value comment as in outcome 1, analysis 1]; P-value calculated using analysis of variance (ANOVA) model with treatment term only in the model

4. Secondary Outcome: Time Weighted Sum of Change From Baseline in the Back Stiffness Score Over 8 Hours
Description: Time weighted sum of change calculated as sum of change from baseline in back stiffness scores from 0 through 8 hours, weighted by time duration between current timepoint and previous timepoint. Based on hourly (from baseline) back stiffness assessment rating from 0 (no muscle stiffness) to 100 (most possible muscle stiffness). Sum of change derived by subtracting score at post-dosing time point from baseline score. Total possible score -800 to 800; higher positive value was indicative of greater improvement.
Time Frame: Baseline (time of wrap application or oral treatment administration) up to 8 hours
Population: ITT population.
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | ThermaCare® | Sham Wrap (Inactive) | Oral Ibuprofen (IBU) | Oral Placebo
Number analyzed (Participants) | 26 | 5 | 5 | 25
scores on a scale | 167.0 (83.7) | 140.6 (71.3) | 105.0 (143.2) | 74.5 (111.3)
Statistical Analysis 1: Comparison: ThermaCare® vs Oral Placebo; Test type: Superiority or Other; p = 0.002, ANOVA — [p-value comment as in outcome 1, analysis 1]; P-value calculated using ANOVA model with treatment term only in the model

5. Secondary Outcome: Time to Treatment Failure
Description: Time to treatment failure defined as time from dosing to the time of rescue medication within the scheduled duration of the study (8 hours); or for participants who withdrew from the study due to lack of efficacy without taking rescue medication, the time of the last assessment was considered the time to treatment failure; or if participant did not take rescue medication, or did not discontinue due to lack of efficacy, the time to treatment failure was considered censored at 8 hours (the scheduled duration of the study).
Time Frame: Baseline (time of wrap application or oral treatment administration) up to 8 hours
Population: ITT population. Time to treatment failure not calculable as there were no treatment failures in this study. No participants required use of rescue medication or discontinued study prior to 8 hour evaluation.
Arm/Group | ThermaCare® | Sham Wrap (Inactive) | Oral Ibuprofen (IBU) | Oral Placebo
Number analyzed (Participants) | 0 | 0 | 0 | 0

6. Secondary Outcome: Individual Time-Point Pain Relief Scores
Description: Pain relief rated hourly (from baseline) by the participant on a 6-point scale: 0=no relief, 1=a little relief, 2=less than half relief, 3=more than half relief, 4=a lot of relief, 5=complete relief.
Time Frame: At 60, 120, 180, 240, 300, 360, 420, and 480 minutes
Population: ITT population.
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | ThermaCare® | Sham Wrap (Inactive) | Oral Ibuprofen (IBU) | Oral Placebo
Number analyzed (Participants) | 26 | 5 | 5 | 25
scores on a scale
  60 minutes | 1.4 (1.1) | 1.0 (0.7) | 1.0 (1.4) | 0.6 (1.1)
  120 minutes | 2.1 (1.1) | 1.6 (1.3) | 1.6 (1.5) | 1.2 (1.3)
  180 minutes | 2.9 (1.2) | 2.2 (1.9) | 2.4 (1.5) | 1.4 (1.4)
  240 minutes | 3.0 (1.2) | 2.2 (1.9) | 2.4 (1.8) | 1.7 (1.5)
  300 minutes | 3.1 (1.2) | 2.0 (2.0) | 2.2 (1.8) | 1.5 (1.5)
  360 minutes | 3.2 (1.2) | 2.4 (1.8) | 2.4 (2.3) | 1.7 (1.5)
  420 minutes | 3.1 (1.4) | 2.0 (2.1) | 2.6 (2.4) | 1.7 (1.6)
  480 minutes | 3.2 (1.4) | 2.2 (1.9) | 2.4 (2.2) | 1.7 (1.5)
Statistical Analysis 1: Comparison: ThermaCare® vs Oral Placebo; 60 minutes timepoint; Test type: Superiority or Other; p = 0.012, ANOVA — [p-value comment as in outcome 1, analysis 1]; P-value from ANOVA model with treatment term only in the model
Statistical Analysis 2: Comparison: ThermaCare® vs Oral Placebo; 120 minutes timepoint; Test type: Superiority or Other; p = 0.016, ANOVA — [p-value comment as in outcome 1, analysis 1]; P-value from ANOVA model with treatment term only in the model
Statistical Analysis 3: Comparison: ThermaCare® vs Oral Placebo; 180 minutes timepoint; Test type: Superiority or Other; p < 0.001, ANOVA — [p-value comment as in outcome 1, analysis 1]; P-value from ANOVA model with treatment term only in the model
Statistical Analysis 4: Comparison: ThermaCare® vs Oral Placebo; 240 minutes timepoint; Test type: Superiority or Other; p = 0.002, ANOVA — [p-value comment as in outcome 1, analysis 1]; P-value from ANOVA model with treatment term only in the model
Statistical Analysis 5: Comparison: ThermaCare® vs Oral Placebo; 300 minutes timepoint; Test type: Superiority or Other; p < 0.001, ANOVA — [p-value comment as in outcome 1, analysis 1]; P-value from ANOVA model with treatment term only in the model
Statistical Analysis 6: Comparison: ThermaCare® vs Oral Placebo; 360 minutes timepoint; Test type: Superiority or Other; p < 0.001, ANOVA — [p-value comment as in outcome 1, analysis 1]; P-value from ANOVA model with treatment term only in the model
Statistical Analysis 7: Comparison: ThermaCare® vs Oral Placebo; 420 minutes timepoint; Test type: Superiority or Other; p = 0.003, ANOVA — [p-value comment as in outcome 1, analysis 1]; P-value from ANOVA model with treatment term only in the model
Statistical Analysis 8: Comparison: ThermaCare® vs Oral Placebo; 480 minutes timepoint; Test type: Superiority or Other; p = 0.001, ANOVA — [p-value comment as in outcome 1, analysis 1]; P-value from ANOVA model with treatment term only in the model

7. Secondary Outcome: Change From Baseline in Individual Time-point Back Stiffness Scores
Description: Low back muscle stiffness rated hourly (from baseline) by the participant by placing a line on a visual analog scale (VAS) from 0 millimeters (mm) to 100 mm in length with 0=no muscle stiffness up to 100 (most possible stiffness).
Time Frame: At 60, 120, 180, 240, 300, 360, 420, and 480 minutes
Population: ITT population.
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | ThermaCare® | Sham Wrap (Inactive) | Oral Ibuprofen (IBU) | Oral Placebo
Number analyzed (Participants) | 26 | 5 | 5 | 25
scores on a scale
  60 minutes | 9.4 (10.8) | 8.4 (10.5) | -3.0 (8.4) | 1.3 (11.8)
  120 minutes | 14.7 (10.4) | 17.6 (10.3) | 8.0 (12.5) | 4.7 (11.5)
  180 minutes | 20.3 (11.8) | 18.6 (12.8) | 14.0 (18.5) | 8.9 (24.2)
  240 minutes | 22.7 (12.2) | 17.6 (12.1) | 18.0 (20.2) | 14.0 (23.2)
  300 minutes | 23.5 (11.8) | 19.2 (11.0) | 18.0 (20.2) | 9.6 (17.4)
  360 minutes | 24.5 (13.1) | 20.8 (10.6) | 18.0 (22.0) | 11.5 (17.8)
  420 minutes | 25.8 (15.7) | 18.0 (10.4) | 18.0 (28.0) | 12.5 (17.1)
  480 minutes | 26.3 (15.8) | 20.4 (10.6) | 14.0 (26.1) | 12.0 (17.1)
Statistical Analysis 1: Comparison: ThermaCare® vs Oral Placebo; 60 minutes timepoint; Test type: Superiority or Other; p = 0.012, ANOVA — [p-value comment as in outcome 1, analysis 1]; P-value from ANOVA model with treatment term only in the model
Statistical Analysis 2: Comparison: ThermaCare® vs Oral Placebo; 120 minutes timepoint; Test type: Superiority or Other; p = 0.002, ANOVA — [p-value comment as in outcome 1, analysis 1]; P-value from ANOVA model with treatment term only in the model
Statistical Analysis 3: Comparison: ThermaCare® vs Oral Placebo; 180 minutes timepoint; Test type: Superiority or Other; p = 0.033, ANOVA — [p-value comment as in outcome 1, analysis 1]; P-value from ANOVA model with treatment term only in the model
Statistical Analysis 4: Comparison: ThermaCare® vs Oral Placebo; 240 minutes timepoint; Test type: Superiority or Other; p = 0.096, ANOVA — [p-value comment as in outcome 1, analysis 1]; P-value from ANOVA model with treatment term only in the model
Statistical Analysis 5: Comparison: ThermaCare® vs Oral Placebo; 300 minutes timepoint; Test type: Superiority or Other; p = 0.002, ANOVA — [p-value comment as in outcome 1, analysis 1]; P-value from ANOVA model with treatment term only in the model
Statistical Analysis 6: Comparison: ThermaCare® vs Oral Placebo; 360 minutes timepoint; Test type: Superiority or Other; p = 0.005, ANOVA — [p-value comment as in outcome 1, analysis 1]; P-value from ANOVA model with treatment term only in the model
Statistical Analysis 7: Comparison: ThermaCare® vs Oral Placebo; 420 minutes timepoint; Test type: Superiority or Other; p = 0.008, ANOVA — [p-value comment as in outcome 1, analysis 1]; P-value from ANOVA model with treatment term only in the model
Statistical Analysis 8: Comparison: ThermaCare® vs Oral Placebo; 480 minutes timepoint; Test type: Superiority or Other; p = 0.004, ANOVA — [p-value comment as in outcome 1, analysis 1]; P-value from ANOVA model with treatment term only in the model

8. Secondary Outcome: Change From Baseline (Bsl) in Combined Flexibility Score: Extension
Description: Flexibility assessed using Paris Plinth table with maximum extension (as if performing a sit-up) of 20 degrees movement. Angle at Bsl and at 4 hours standardized to 100 for assessment of maximum angle (x degrees), x degrees minus 5, and x degrees plus 5. Flexibility score derived using standardized value and VAS score (participant rating of pain by marking level of pain on 100 mm line 0=no pain up to 100=worst pain). Final derived data for extension flexibility were average of the extension flexibility data on the combined score (range -66 to 552); higher value indicated greater improvement.
Time Frame: Baseline (time of wrap application or oral treatment administration) and 4 hours
Population: ITT population.
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | ThermaCare® | Sham Wrap (Inactive) | Oral Ibuprofen (IBU) | Oral Placebo
Number analyzed (Participants) | 26 | 5 | 5 | 25
scores on a scale
  At Maximum degrees | 13.7 (34.8) | -4.1 (35.6) | 12.7 (23.1) | 4.3 (23.3)
  At Minus 5 degrees | 17.7 (39.1) | 8.4 (43.2) | 8.0 (39.7) | 39.0 (133.6)
  At Plus 5 degrees (beyond maximum) | 15.8 (36.4) | -5.8 (31.6) | 9.3 (30.9) | 1.5 (17.7)
Statistical Analysis 1: Comparison: ThermaCare® vs Oral Placebo; At Maximum degrees; Test type: Superiority or Other; p = 0.268, ANOVA — [p-value comment as in outcome 1, analysis 1]; P-value from ANOVA model with treatment term only in the model
Statistical Analysis 2: Comparison: ThermaCare® vs Oral Placebo; At Minus 5 degrees; Test type: Superiority or Other; p = 0.419, ANOVA — [p-value comment as in outcome 1, analysis 1]; P-value from ANOVA model with treatment term only in the model
Statistical Analysis 3: Comparison: ThermaCare® vs Oral Placebo; At Plus 5 degrees (beyond maximum); Test type: Superiority or Other; p = 0.086, ANOVA — [p-value comment as in outcome 1, analysis 1]; P-value from ANOVA model with treatment term only in the model

9. Secondary Outcome: Change From Baseline (Bsl) in Overall Combined Flexibility Score: Side-to-Side
Description: Flexibility assessed using Paris Plinth table with maximum side-to-side movement of plus or minus (+/-) 10 degrees for left, and right (L, R), movement. Angle at Bsl and 4 hours standardized to 100 for assessment of maximum angle (x degrees), x degrees - 5, and x degrees + 5. Flexibility score derived using standardized value and VAS score (participant rating of level of pain on 100 mm line 0=no pain to 100=worst pain). Final derived data for overall flexibility was the average of side-to-side (L, R) flexibility data on the combined score (range -81 to 264); higher value=greater improvement.
Time Frame: Baseline (time of wrap application or oral treatment administration) and 4 hours
Population: ITT population.
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | ThermaCare® | Sham Wrap (Inactive) | Oral Ibuprofen (IBU) | Oral Placebo
Number analyzed (Participants) | 26 | 5 | 5 | 25
scores on a scale
  At Maximum degrees | 13.9 (28.7) | 14.0 (27.2) | 3.8 (21.6) | 0.7 (21.7)
  At Minus 5 degrees | 9.5 (37.3) | 2.3 (2.8) | -18.0 (38.0) | 14.2 (65.5)
  At Plus 5 degrees (beyond maximum) | 11.0 (32.5) | 14.8 (31.3) | 10.9 (25.1) | 2.0 (14.5)
Statistical Analysis 1: Comparison: ThermaCare® vs Oral Placebo; At Maximum degrees; Test type: Superiority or Other; p = 0.067, ANOVA — [p-value comment as in outcome 1, analysis 1]; P-value from ANOVA model with treatment term only in the model
Statistical Analysis 2: Comparison: ThermaCare® vs Oral Placebo; At Minus 5 degrees; Test type: Superiority or Other; p = 0.757, ANOVA — [p-value comment as in outcome 1, analysis 1]; P-value from ANOVA model with treatment term only in the model
Statistical Analysis 3: Comparison: ThermaCare® vs Oral Placebo; At Plus 5 degrees (beyond maximum); Test type: Superiority or Other; p = 0.219, ANOVA — [p-value comment as in outcome 1, analysis 1]; P-value from ANOVA model with treatment term only in the model

10. Secondary Outcome: Change From Baseline (Bsl) in Overall Combined Flexibility Score: Rotation
Description: Flexibility assessed using Paris Plinth table with maximum rotation at waist of plus or minus (+/-) 30 degrees for left, and right (L, R), movement. Angle at Bsl and at 4 hours standardized to 100 for assessment of maximum angle (x degrees), x degrees - 5, and x degrees + 5. Flexibility score derived using standardized value and VAS score (participant rating of level of pain on 100 mm line 0=no pain up to 100=worst pain). Final derived data for overall flexibility were the average of rotation (L, R) flexibility data on combined score (range -80 to 155); higher value=greater improvement.
Time Frame: Baseline (time of wrap application or oral treatment administration) and 4 hours
Population: ITT population.
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | ThermaCare® | Sham Wrap (Inactive) | Oral Ibuprofen (IBU) | Oral Placebo
Number analyzed (Participants) | 26 | 5 | 5 | 25
scores on a scale
  At Maximum degrees | 9.9 (19.0) | 24.1 (12.5) | 12.1 (18.5) | -0.2 (16.4)
  At Minus 5 degrees | 13.0 (33.3) | 35.9 (22.0) | 6.8 (21.5) | 4.1 (42.9)
  At Plus 5 degrees (beyond maximum) | 10.0 (22.2) | 33.4 (27.2) | 14.5 (19.8) | -1.4 (13.9)
Statistical Analysis 1: Comparison: ThermaCare® vs Oral Placebo; At Maximum degrees; Test type: Superiority or Other; p = 0.043, ANOVA — [p-value comment as in outcome 1, analysis 1]; P-value from ANOVA model with treatment term only in the model
Statistical Analysis 2: Comparison: ThermaCare® vs Oral Placebo; At Minus 5 degrees; Test type: Superiority or Other; p = 0.388, ANOVA — [p-value comment as in outcome 1, analysis 1]; P-value from ANOVA model with treatment term only in the model
Statistical Analysis 3: Comparison: ThermaCare® vs Oral Placebo; At Plus 5 degrees (beyond maximum); Test type: Superiority or Other; p = 0.039, ANOVA — [p-value comment as in outcome 1, analysis 1]; P-value from ANOVA model with treatment term only in the model

11. Secondary Outcome: Change From Baseline in the Angle Measurement at Maximum Flexion for Flexibility Measures: Extension
Description: Participant placed in a prone position on Paris Plinth table which is moved at 1 degree per second to maximum movement of 20 degrees for extension (as if performing a sit-up) to the degree of movement at which participant perceives discomfort or pain. Higher score indicated greater improvement.
Time Frame: Baseline (time of wrap application or oral treatment administration) and 4 hours
Population: ITT population.
Measure: Mean (Standard Deviation); unit: degrees
Arm/Group | ThermaCare® | Sham Wrap (Inactive) | Oral Ibuprofen (IBU) | Oral Placebo
Number analyzed (Participants) | 26 | 5 | 5 | 25
degrees | 1.4 (3.0) | -1.1 (3.1) | 0.5 (2.9) | 1.2 (4.6)
Statistical Analysis 1: Comparison: ThermaCare® vs Oral Placebo; Test type: Superiority or Other; p = 0.797, ANOVA — [p-value comment as in outcome 1, analysis 1]; P-value from ANOVA model with treatment term only in the model

12. Secondary Outcome: Change From Baseline in the Angle Measurement at Maximum Flexion for Flexibility Measures: Side-to-Side
Description: Participant placed in a prone position on Paris Plinth table which is moved at 1 degree per second to maximum movement +/- 10 degrees for left, and right, side-to-side movement to the degree of movement at which participant perceives discomfort or pain. Maximum flexion based on the average of the left and right side-to-side scores. Higher score indicated greater improvement.
Time Frame: Baseline (time of wrap application or oral treatment administration) and 4 hours
Population: ITT population.
Measure: Mean (Standard Deviation); unit: degrees
Arm/Group | ThermaCare® | Sham Wrap (Inactive) | Oral Ibuprofen (IBU) | Oral Placebo
Number analyzed (Participants) | 26 | 5 | 5 | 25
degrees | 0.1 (1.2) | 0.4 (1.0) | -0.3 (0.4) | -0.2 (1.4)
Statistical Analysis 1: Comparison: ThermaCare® vs Oral Placebo; Test type: Superiority or Other; p = 0.371, ANOVA — [p-value comment as in outcome 1, analysis 1]; P-value from ANOVA model with treatment term only in the model

13. Secondary Outcome: Change From Baseline in the Angle Measurement at Maximum Flexion for Flexibility Measures: Rotation
Description: Participant placed in a prone position on Paris Plinth table which is moved at 1 degree per second to maximum rotation at waist of +/- 30 degrees for left, and right, movement to the degree of movement at which participant perceives discomfort or pain. Maximum flexion based on the average of the left and right rotation scores. Higher score indicated greater improvement.
Time Frame: Baseline (time of wrap application or oral treatment administration) and 4 hours
Population: ITT population.
Measure: Mean (Standard Deviation); unit: degrees
Arm/Group | ThermaCare® | Sham Wrap (Inactive) | Oral Ibuprofen (IBU) | Oral Placebo
Number analyzed (Participants) | 26 | 5 | 5 | 25
degrees | 0.6 (2.5) | 1.3 (1.4) | -0.6 (0.6) | -0.6 (3.3)
Statistical Analysis 1: Comparison: ThermaCare® vs Oral Placebo; Test type: Superiority or Other; p = 0.122, ANOVA — [p-value comment as in outcome 1, analysis 1]; P-value from ANOVA model with treatment term only in the model

14. Secondary Outcome: Change From Baseline (Bsl) in Pain Measurement for Flexibility Measure: Extension
Description: Flexibility assessed using Paris Plinth table with maximum extension of 20 degrees movement (as if performing a sit-up). When participant feels discomfort or pain, participant places a mark to rate discomfort/pain (maximum) on a VAS of 100 mm in length with 0=no discomfort/no pain up to 100=most discomfort/most pain. Movement decreased 5 degrees (minus) and discomfort rated on VAS. Movement increased 5 degrees (plus) beyond first point when pain was reported and discomfort/pain again rated on the VAS. Higher score indicated greater discomfort/pain.
Time Frame: Baseline (time of wrap application or oral treatment administration) and 4 hours
Population: ITT population.
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | ThermaCare® | Sham Wrap (Inactive) | Oral Ibuprofen (IBU) | Oral Placebo
Number analyzed (Participants) | 26 | 5 | 5 | 25
scores on a scale
  At Maximum degrees | 4.7 (25.0) | -0.8 (32.9) | 10.4 (15.4) | -0.6 (11.0)
  At Minus 5 degrees | 2.7 (15.1) | 7.4 (24.7) | 7.2 (23.3) | -1.8 (17.8)
  At Plus 5 degrees (beyond maximum) | 9.5 (24.7) | -5.6 (32.1) | 12.6 (30.7) | 2.0 (11.5)
Statistical Analysis 1: Comparison: ThermaCare® vs Oral Placebo; At Maximum degrees; Test type: Superiority or Other; p = 0.355, ANOVA — [p-value comment as in outcome 1, analysis 1]; P-value from ANOVA model with treatment term only in the model
Statistical Analysis 2: Comparison: ThermaCare® vs Oral Placebo; At Minus 5 degrees; Test type: Superiority or Other; p = 0.371, ANOVA — [p-value comment as in outcome 1, analysis 1]; P-value from ANOVA model with treatment term only in the model
Statistical Analysis 3: Comparison: ThermaCare® vs Oral Placebo; At Plus 5 degrees (beyond maximum); Test type: Superiority or Other; p = 0.216, ANOVA — [p-value comment as in outcome 1, analysis 1]; P-values from ANOVA model with treatment treatment term only in the model

15. Secondary Outcome: Change From Baseline in Pain Measurement for Flexibility Measure: Side-to-Side
Description: Flexibility assessed using Paris Plinth table with maximum side-to-side movement of +/- 10 degrees for L, R movement. When participant feels discomfort or pain, participant places a mark to rate discomfort/pain (maximum) on a VAS of 100 mm in length with 0=no discomfort/no pain up to 100=most discomfort/most pain. Movement decreased 5 degrees (minus) and discomfort rated on VAS. Movement increased 5 degrees (plus) beyond first point when pain was reported and discomfort/pain again rated on the VAS. Analyses based on the average of L, R scores. Higher score indicated greater discomfort/pain.
Time Frame: Baseline (time of wrap application or oral treatment administration) and 4 hours
Population: ITT population.
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | ThermaCare® | Sham Wrap (Inactive) | Oral Ibuprofen (IBU) | Oral Placebo
Number analyzed (Participants) | 26 | 5 | 5 | 25
scores on a scale
  At Maximum degrees | 7.9 (13.4) | 5.0 (10.9) | 6.6 (21.2) | -0.3 (15.4)
  At Minus 5 degrees | 4.2 (10.7) | 4.6 (5.8) | 2.2 (18.3) | 2.6 (10.4)
  At Plus 5 degrees (beyond maximum) | 5.9 (18.1) | 7.3 (16.0) | 11.2 (25.4) | 0.9 (12.7)
Statistical Analysis 1: Comparison: ThermaCare® vs Oral Placebo; At Maximum degrees; Test type: Superiority or Other; p = 0.054, ANOVA — [p-value comment as in outcome 1, analysis 1]; P-value from ANOVA model with treatment term only in the model
Statistical Analysis 2: Comparison: ThermaCare® vs Oral Placebo; At Minus 5 degrees; Test type: Superiority or Other; p = 0.600, ANOVA — [p-value comment as in outcome 1, analysis 1]; P-value from ANOVA model with treatment term only in the model
Statistical Analysis 3: Comparison: ThermaCare® vs Oral Placebo; At Plus 5 degrees (beyond maximum); Test type: Superiority or Other; p = 0.294, ANOVA — [p-value comment as in outcome 1, analysis 1]; P-value from ANOVA model with treatment term only in the model

16. Secondary Outcome: Change From Baseline in Pain Measurement for Flexibility Measure: Rotation
Description: Flexibility assessed using Paris Plinth table with maximum rotation at waist of +/- 30 degrees for L, R movement. When participant feels discomfort or pain, participant places a mark to rate discomfort/pain (maximum) on a VAS of 100 mm in length with 0=no discomfort/no pain up to 100=most discomfort/most pain. Movement decreased 5 degrees (minus) and discomfort rated on VAS. Movement increased 5 degrees (plus) beyond first point when pain was reported and discomfort/pain again rated on the VAS. Analyses based on the average of L, R scores. Higher score indicated greater discomfort/pain.
Time Frame: Baseline (time of wrap application or oral treatment administration) and 4 hours
Population: ITT population.
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | ThermaCare® | Sham Wrap (Inactive) | Oral Ibuprofen (IBU) | Oral Placebo
Number analyzed (Participants) | 26 | 5 | 5 | 25
scores on a scale
  At Maximum degrees | 7.4 (15.9) | 17.4 (9.0) | 15.7 (18.9) | 0.2 (13.5)
  At Minus 5 degrees | 5.4 (17.8) | 19.4 (8.4) | 12.5 (15.6) | 3.2 (13.5)
  At Plus 5 degrees (beyond maximum) | 9.3 (21.5) | 25.4 (14.1) | 20.9 (18.1) | -1.2 (12.0)
Statistical Analysis 1: Comparison: ThermaCare® vs Oral Placebo; At Maximum degrees; Test type: Superiority or Other; p = 0.088, ANOVA — [p-value comment as in outcome 1, analysis 1]; P-value from ANOVA model with treatment term only in the model
Statistical Analysis 2: Comparison: ThermaCare® vs Oral Placebo; At Minus 5 degrees; Test type: Superiority or Other; p = 0.625, ANOVA — [p-value comment as in outcome 1, analysis 1]; P-value from ANOVA model with treatment term only in the model
Statistical Analysis 3: Comparison: ThermaCare® vs Oral Placebo; At Plus 5 degrees (beyond maximum); Test type: Superiority or Other; p = 0.034, ANOVA — [p-value comment as in outcome 1, analysis 1]; P-value from ANOVA model with treatment term only in the model

17. Secondary Outcome: Number of Participants Per Categorical Score for Global Assessment of Study Treatment
Description: At hour 8, or at the time of rescue, if it occurred, participants performed a global assessment in their diary in response to the question: How would you rate the study treatment as a pain reliever? Very Poor=0, Poor=1, Fair=2, Good=3, Very Good=4, Excellent=5.
Time Frame: Baseline (time of wrap application or oral treatment administration) up to 8 hours
Population: ITT population.
Measure: Number; unit: participants
Arm/Group | ThermaCare® | Sham Wrap (Inactive) | Oral Ibuprofen (IBU) | Oral Placebo
Number analyzed (Participants) | 26 | 5 | 5 | 25
participants
  Very poor=0 | 0 | 1 | 0 | 6
  Poor=1 | 0 | 0 | 1 | 5
  Fair=2 | 4 | 0 | 1 | 10
  Good=3 | 10 | 2 | 2 | 1
  Very good=4 | 9 | 0 | 1 | 1
  Excellent=5 | 2 | 0 | 0 | 2
  Response missing | 1 | 2 | 0 | 0
Statistical Analysis 1: Comparison: ThermaCare® vs Oral Placebo; Test type: Superiority or Other; p < 0.001, Cochran-Mantel-Haenszel — [p-value comment as in outcome 1, analysis 1]; P-value from the Cochran-Mantel-Haenszel test with modified ridit scores

ADVERSE EVENTS:
Time Frame: Baseline up to 5 days after the 8 hour evaluation period.
Description: The same event may appear as both an AE and a SAE. However, what is presented are distinct events. An event may be categorized as serious in one subject and as nonserious in another subject, or one subject may have experienced both a serious and nonserious event during the study.
Arm/Group | ThermaCare® | Sham Wrap (Inactive) | Oral Ibuprofen (IBU) | Oral Placebo
Serious Adverse Events (participants affected / at risk) | 0/26 | 0/5 | 0/5 | 0/25
Other Adverse Events (participants affected / at risk) | 2/26 | 0/5 | 0/5 | 0/25
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | ThermaCare® (N=26) | Sham Wrap (Inactive) (N=5) | Oral Ibuprofen (IBU) (N=5) | Oral Placebo (N=25)
Headache (Nervous system disorders) | 2 | 0 | 0 | 0
Asthma (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0

LIMITATIONS AND CAVEATS:
No primary endpoint was prespecified in this Pilot study; 1 key efficacy endpoint was selected for reporting purposes only.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Pfizer has the right to review disclosures, requesting a delay of less than 60 days. Investigator will postpone single center publications until after the disclosure of pooled data (all sites), less than 12 months from study completion/termination at all participating sites. Investigator may not disclose previously undisclosed confidential information other than study results.